CLINICAL TRIAL: NCT03950011
Title: Database for Data Collection in the Context of an Enhanced Recovery After Surgery Program in Oncology Surgery
Acronym: BDD RAAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BDD RAAC-IPC 2016-011; 2174848 (Other: CNIL)
Record Dates: First submitted 2018-09-20; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Oncology
Keywords: Enhanced Recovery After Surgery Program (ERP)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERP: Any patient requiring oncologic surgery, including hysterectomy or curettage, posterior pelvectomy, conventional laparoscopic or assisted robotic surgery, or laparotomy for cervical or cervical cancer or ovarian cancer, body or cervix uterus and ovaries as well as benign pathologies or borderline malignancy.
  Interventions: Procedure: Enhanced recovery after surgery program

INTERVENTIONS:
Procedure: Enhanced recovery after surgery program — Enhanced Recovery After Surgery Programs (ERP) includes multimodal approaches of perioperative patient's clinical pathways designed to achieve early recovery after surgery and a decreased length of hospital stay (LOS).

SUMMARY:
Enhanced Recovery After Surgery Programs (ERP) includes multimodal approaches of perioperative patient's clinical pathways designed to achieve early recovery after surgery and a decreased length of hospital stay (LOS).

DETAILED DESCRIPTION:
This database would also allow an objective evaluation of the quality of the surgical management and the follow-up.

One of the evaluation criteria will be measured by the quantity and quality of publications from this database, and also by the increase in the activity of the service concerned.

ELIGIBILITY:
Inclusion Criteria:

* Any patient operated including hysterectomy and or curettage, posterior pelvectomy, conventional laparoscopic or assisted robot, or laparotomy at the Paoli-Calmettes Institute from 01 2016 to 12 2017, and incrementation from 2018.

Exclusion Criteria:

* Non applicable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — uterine or cervical cancer or ovarian cancer
Study Population: Any patient operated including hysterectomy and or curettage, posterior pelvectomy, conventional laparoscopic or assisted robot, or laparotomy at the Paoli-Calmettes Institute from 01 2016 to 12 2017, and incrementation from 2018.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Data collection | 4 years
  Restrospective and prospective data collection

SECONDARY OUTCOMES:
Evaluation of the quality of surgical management | 4 days
  characteristics of the surgery according to the type of diagnosis
Post-operative complications | 4 days
  post-operative complications in hospitalization and post-operative complications after leaving hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

REFERENCES:
- [Result] Lambaudie E, de Nonneville A, Brun C, Laplane C, N'Guyen Duong L, Boher JM, Jauffret C, Blache G, Knight S, Cini E, Houvenaeghel G, Blache JL. Enhanced recovery after surgery program in Gynaecologic Oncological surgery in a minimally invasive techniques expert center. BMC Surg. 2017 Dec 28;17(1):136. doi: 10.1186/s12893-017-0332-9. PMID 29282059